CLINICAL TRIAL: NCT04190407
Title: Intravenous Access Time With the Corresponding Bispectral Index Value During Anesthesia Induction in Pediatric Patients
Brief Title: Intravenous Access Time in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Zeynep Nur Orhon, Principal Investigator, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IstanbulMUzeynep1
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Intravenous Access; Pediatric Patient
Keywords: Intravenous access; Sevoflurane; Bispectral index; Pediatric patient

STUDY DESIGN:
Intervention Model Description: Patients with American Society of Anesthesiologists physical status I or II; age between 2 months to 11 years; and scheduled for day case surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients scheduled for day case surgery (Other): A tourniquet was used to raise the vein for entry into the vein every 15 s after the ciliary reflex disappeared. If the patient showed no response to the tourniquet (movement, coughing, or laryngospasm), an experienced anesthesiologist entered a vein in the dorsum of one hand using a 22-24 gauge cannula.
  Interventions: Behavioral: Intravenous access

INTERVENTIONS:
Behavioral: Intravenous access — A tourniquet was used to raise the vein for entry into the vein every 15 s after the ciliary reflex disappeared. If the patient showed no response to the tourniquet (movement, coughing, or laryngospasm), an experienced anesthesiologist entered a vein in the dorsum of one hand using a 22-24 gauge cannula.

SUMMARY:
In pediatric patients with no vascular access, anesthesia induction is usually achieved with sevoflurane. The aim of investigators to evaluate the optimum intravenous access time and the corresponding bispectral index (BIS) value in pediatric surgery under sevoflurane anesthesia.

DETAILED DESCRIPTION:
Patients undergoing anesthesia induction must have at least one vascular access opened for administration of intravenous drugs and fluid. In pediatric patients, fear of needles and anxiety about pain can cause discomfort. For this reason, inhalational anesthetics are commonly used for anesthesia induction in children. An ideal inhalational anesthetic agent should have a smooth and fast onset, little irritation to the respiratory tract, and no undesirable side effects. Sevoflurane meets almost all these criteria, so it is commonly used for anesthesia induction in pediatric patients.

Studies related to the induction of anesthesia with sevoflurane have mostly focused on the ease of LMA insertion, the recovery characteristics, the hemodynamic variabilities, comparison of high and low initial sevoflurane concentrations, and cost comparisons between fixed 8% versus incremental techniques. However, after loss of consciousness, children subjected to early intravenous cannulation during sevoflurane induction can display movement, breath holding, coughing, and even laryngospasm. Only limited data are available in the literature regarding intravenous access time at anesthesia induction. The aim of the present study was to evaluate the bispectral index (BIS) values and sevoflurane concentrations during induction of anesthesia and to determine the optimum intravenous access time in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I or II
* Age between 2 months to 11 years
* Patients scheduled for day case surgery (including inguinoscrotal hernia or hydrocele, undescended testis, hypospadias, or routine circumcision)
* Diagnostic procedures (e.g., cystoscopy) or external ventricular drainage.

Exclusion Criteria:

* Obesity
* Malnutrition
* Gastroesophageal reflux disease
* Allergy
* Sensitivity to volatile anesthetics
* Procedures lasting more than two hours.

Ages: 2 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Intravenous access time with the corresponding bispectral index value during anesthesia induction in pediatric patients | 12 months
  It was evaluated the optimum intravenous access time and the corresponding bispectral index (BIS) value in pediatric surgery under sevoflurane anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep N Orhon, Dr., Principal Investigator — Istanbul Medeniyet University

IPD SHARING:
Plan to Share IPD: No